CLINICAL TRIAL: NCT03250377
Title: An Open-Label, Multicenter, Follow-up Study to Evaluate the Long-Term Safety and Efficacy of Brivaracetam Used as Adjunctive Treatment in Subjects >=16 Years of Age With Partial Seizures With or Without Secondary Generalization
Brief Title: A Study to Test the Safety/ Efficacy of Brivaracetam (BRV) Used as Adjunctive Treatment in Subjects >=16 Years of Age With Partial Seizures With or Without Secondary Generalization
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP0085
Record Dates: First submitted 2017-07-31; First posted 2017-08-15 (Actual); Results first posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Partial Seizures With or Without Secondary Generalization; Epilepsy
Keywords: Brivaracetam; Epilepsy; Partial seizures with or without secondary generalization; Briviact
MeSH Terms: conditions — Epilepsy | interventions — brivaracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brivaracetam (Experimental): Subjects randomized to this arm will receive open-label Brivaracetam
  Interventions: Drug: Brivaracetam

INTERVENTIONS:
Drug: Brivaracetam — * Pharmaceutical form: Film-coated tablet
  * Concentration: 25 mg and 50 mg
  * Route of administration: Oral use
  Other Names: Briviact

SUMMARY:
The purpose of the study is to evaluate the long-term safety and tolerability of Brivaracetam (BRV) in focal epilepsy subjects with partial seizures and to evaluate the maintenance of efficacy of BRV over time.

ELIGIBILITY:
Inclusion Criteria:

* Male/female study participant from 16 years of age or older. Study participant who are not legal adults may only be included where legally permitted and ethically accepted
* Study participant completed the Treatment Period and Transition Period of EP0083 or is ongoing in N01379 sites in Japan
* Female study participants with childbearing potential are eligible if they use a medically accepted contraceptive method
* Inclusion Criteria for directly enrollers only: Study participant has 1 to <8 partial seizures (according to the 1981 International League Against Epilepsy (ILAE) classification) during the 8 weeks prior to brivaracetam (BRV) administration

Exclusion Criteria:

* Study participant has developed hypersensitivity to any components of the investigational medicinal product (IMP) or comparative drugs as stated in this protocol during the course of the core study
* Severe medical, neurological or psychiatric disorders, or laboratory values which may have an impact on the safety of the study participant
* Poor compliance with the visit schedule or medication intake in the previous BRV studies
* Planned participation in any other clinical study of another investigational drug or device during this study
* Pregnant or lactating woman
* Any medical condition which, in the Investigator's opinion, warrants exclusion
* Study participant has a lifetime history of suicide attempt or has suicidal ideation in the past 6 months
* Study participant has >2 x upper limit of normal (ULN) of any of the following at the Entry Visit (EV): alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), or >ULN total bilirubin (≥1.5x ULN total bilirubin if known Gilbert's syndrome)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2017-08-05 (Actual); Primary Completion 2024-12-24 (Actual); Study Completion 2024-12-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (59):
- China (19):
  - Ep0085 905, Beijing
  - Ep0085 901, Chengdu
  - Ep0085 902, Guangzhou
  - Ep0085 909, Guangzhou
  - Ep0085 917, Guangzhou
  - Ep0085 920, Guangzhou
  - Ep0085 924, Guangzhou
  - Ep0085 912, Hangzhou
  - Ep0085 908, Lanzhou
  - Ep0085 921, Nanchang
  - Ep0085 926, Pingxiang
  - Ep0085 910, Shijiazhuang
  - Ep0085 925, Suzhou
  - Ep0085 913, Wenzhou
  - Ep0085 930, Xinxiang
  - Ep0085 916, Yinchuan
  - Ep0085 918, Zhanjiang
  - Ep0085 904, Zhengzhou
  - Ep0085 923, Zunyi
- Japan (40):
  - Ep0085 148, Adachi-ku
  - Ep0085 116, Asaka
  - Ep0085 126, Bunkyō City
  - Ep0085 127, Bunkyō City
  - Ep0085 122, Hachinohe
  - Ep0085 111, Hamamatsu
  - Ep0085 141, Higashisonogi-gun Kawatana-cho
  - Ep0085 110, Hiroshima
  - Ep0085 121, Itami
  - Ep0085 102, Kagoshima
  - Ep0085 142, Kamakura
  - Ep0085 140, Kawasaki
  - Ep0085 123, Kodaira
  - Ep0085 115, Kokubunji
  - Ep0085 132, Kōriyama
  - Ep0085 112, Kōshi
  - Ep0085 128, Kurume
  - Ep0085 124, Kyoto
  - Ep0085 147, Kyoto
  - Ep0085 105, Nagakute
  - Ep0085 118, Nagoya
  - Ep0085 136, Nagoya
  - Ep0085 117, Nara
  - Ep0085 129, Neyagawa
  - Ep0085 106, Niigata
  - Ep0085 850, Osaka
  - Ep0085 130, Ôsaka
  - Ep0085 131, Ōtsu
  - Ep0085 114, Saitama
  - Ep0085 101, Sapporo
  - Ep0085 103, Sendai
  - Ep0085 144, Shinjuku-ku
  - Ep0085 104, Shizuoka
  - Ep0085 108, Suita
  - Ep0085 137, Suita
  - Ep0085 138, Tsukuba
  - Ep0085 133, Ushiku
  - Ep0085 109, Yamagata
  - Ep0085 120, Yokohama
  - Ep0085 150, Yokohama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fujimoto A, Qin B, Bourikas D, Dickson N, Moseley B, Sano T, Soma T, Sun W, Watanabe J, Zhou D, Inoue Y. Safety, Tolerability, and Efficacy of Adjunctive Brivaracetam in Japanese and Chinese Patients with Focal-Onset Seizures: Interim Analysis of a Phase 3 Open-Label Extension Trial. Adv Ther. 2025 Sep;42(9):4335-4349. doi: 10.1007/s12325-025-03253-0. Epub 2025 Jun 23. PMID 40549270

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in August 2017 and concluded in December 2024.
Pre-assignment Details: The Participant Flow refers to the Safety Set (SS). Study consisted of the Evaluation period (duration for rollover participants - 84 Months and for direct enrollers - 39 Months); Down-titration period (4 weeks); drug-free period (2 weeks).
Groups:
- EP0083 Placebo: Participants who received Placebo in study EP0083 (NCT03083665) and completed the Treatment and Transition Period of study EP0083 are rolled over to this study and received brivaracetam (BRV) 50 milligram per day (mg/day) two times (bid) (in total 100 mg/day) at Visit 1 (study entry) and were maintained at this dose for at least 2 weeks unless the participant was unable to tolerate treatment during evaluation period (from Visit 1 to end of study visit or early discontinuation visit i.e. up to 84 months). Upon completion or early discontinuation from EP0085, there was a Down-Titration Period of 4 weeks to decrease in dose in steps on a weekly basis, up to 25 mg/day, followed by a 2-week Study Drug-Free Period during which the participant did not receive study drug. The BRV dose was adjusted (based on the individual participants' s seizure control and tolerability) between 50 mg/day and 200 mg/day during the study.
- EP0083 BRV All: Participants rolled over from study EP0083 received BRV 50 mg/day bid (in total 100 mg/day) at Visit 1 (study entry) and were maintained at this dose for at least 2 weeks unless the participant was unable to tolerate treatment during evaluation period (from Visit 1 to end of study visit or early discontinuation visit i.e. up to 84 months). Upon completion or early discontinuation from EP0085, there was a Down-Titration Period of 4 weeks to decrease in dose in steps on a weekly basis, up to 25 mg/day, followed by a 2-week Study Drug-Free Period during which the participant did not receive study drug. The BRV dose was adjusted (based on the individual participants' s seizure control and tolerability) between 50 mg/day and 200 mg/day during the study.
- N01379 BRV: Participants rolled over from study N01379 (NCT01339559) (core study N01358 [NCT01261325]) received BRV 200 mg/day during the evaluation period (from Visit 1 to end of study visit or early discontinuation visit i.e. up to 84 months). Upon completion or early discontinuation from EP0085, there was a Down-Titration Period of 4 weeks to decrease in dose in steps on a weekly basis, up to 25 mg/day, followed by a 2-week Study Drug-Free Period during which the participant did not receive study drug. The BRV dose was adjusted (based on the individual participants' s seizure control and tolerability) between 50 mg/day and 200 mg/day during the study.
- Direct Enrollers BRV: Participants directly enrolled in this study received BRV 50mg bid (in total 100 mg/day) at Visit 1 (study entry) and were maintained at this dose for at least 2 weeks unless the participant was unable to tolerate treatment during evaluation period (from Visit 1 to end of study visit or early discontinuation visit i.e. Up to 84 Month, however, were evaluated for 39 months only due to late enrollment). Upon completion or early discontinuation from EP0085, there was a Down-Titration Period of 4 weeks to decrease in dose in steps on a weekly basis, up to 25 mg/day, followed by a 2-week Study Drug-Free Period during which the participant did not receive study drug. The BRV dose was adjusted (based on the individual participants' s seizure control and tolerability) between 50 mg/day and 200 mg/day during the study.
Period: Overall Study
Arm/Group | EP0083 Placebo | EP0083 BRV All | N01379 BRV | Direct Enrollers BRV
Started | 54 | 112 | 7 | 34
Evaluation Period (Participants who entered Visit 1 of EP0085 were considered starting the Evaluation Period.) | 54 | 112 | 7 | 34
Down-Titration Period (Participants who had an Early Discontinuation Visit (EDV) and had at least 1 dose of study drug after the date of EDV were considered to start Down-Titration Period.) | 20 | 32 | 5 | 15
Study Drug-Free Period (Participants who had at least one contact after the date of the last dose of BRV were considered to start study Drug-Free period.) | 39 | 76 | 5 | 17
Completed | 37 | 74 | 4 | 20
Not Completed | 17 | 38 | 3 | 14
Not completed — Adverse Event | 2 | 4 | 0 | 4
Not completed — Lack of Efficacy | 5 | 14 | 1 | 3
Not completed — Protocol Violation | 0 | 2 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 7 | 0 | 4
Not completed — Investigator's Judgment | 1 | 0 | 0 | 0
Not completed — She wanted to change other therapeutic medication | 1 | 0 | 0 | 0
Not completed — The Subject Go Abroad and Not Return | 1 | 0 | 0 | 0
Not completed — Epilepsy Surgery | 0 | 1 | 2 | 0
Not completed — Subject moved to kanagawa (faraway from clinic) | 0 | 1 | 0 | 0
Not completed — Request From The Sponsor | 0 | 1 | 0 | 0
Not completed — Subject did not follow procedure or study drug | 0 | 1 | 0 | 0
Not completed — Subject stopped drug; did not wish to continue | 0 | 1 | 0 | 0
Not completed — Subjects did not follow procedures or medication | 0 | 1 | 0 | 0
Not completed — Pregnancy Event | 0 | 1 | 0 | 0
Not completed — PI's opinion:Subject noncompliant with medication | 0 | 1 | 0 | 0
Not completed — Subjects felt no effect;want to discontinue study | 0 | 1 | 0 | 0
Not completed — Subjects underweight; intolerant to study drugs | 0 | 1 | 0 | 0
Not completed — Patient requested to change hospital | 0 | 0 | 0 | 1
Not completed — Admission To Geriatric Health Facility | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set (SS) which consisted of all participants who took at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | EP0083 Placebo | EP0083 BRV All | N01379 BRV | Direct Enrollers BRV | Total
Number analyzed (Participants) | 54 | 112 | 7 | 34 | 207
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (11.6) | 35.8 (13.5) | 40.7 (10.9) | 42.2 (18.6) | 36.7 (14.1)
Age, Customized [Count of Participants; unit: Participants]
  12 - <18 yrs | 2 | 4 | 0 | 1 | 7
  18 - <65 yrs | 52 | 104 | 7 | 29 | 192
  65 - <85 yrs | 0 | 4 | 0 | 3 | 7
  >=85 yrs | 0 | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 53 | 3 | 19 | 107
  Male | 22 | 59 | 4 | 15 | 100
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 54 | 112 | 7 | 34 | 207
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 32 | 58 | 7 | 34 | 131
  Chinese | 22 | 53 | 0 | 0 | 75
  Other | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. Treatment-emergent AEs (TEAEs) were defined as AEs that had onset on or after the day of first BRV dose in EP0085 study.
Time Frame: From Baseline until end of the safety follow up (up to 88.5 months)
Population: The Safety Set consisted of all participants who took at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | EP0083 Placebo | EP0083 BRV All | N01379 BRV | Direct Enrollers BRV
Number analyzed (Participants) | 54 | 112 | 7 | 34
percentage of participants | 88.9 | 95.5 | 100 | 94.1

2. Secondary Outcome: Percent Change in Partial Seizure Frequency (PSF) Per 28 Days From Baseline of EP0083 or N01358 to the Evaluation Period for Rollover Study Participants
Description: The seizure frequency was calculated as number of seizures per 28 days. Percent change of 28 day PSF from Baseline was defined as the percentage reduction of 28 day PSF for a designated post-baseline period in EP0085 compared with the Baseline 28 day PSF in the core study. Change in seizure frequency from Baseline was calculated: percent change = ([Baseline 28 day PSF - Post Baseline 28 day PSF]/[Baseline 28 day PSF]) × 100. For rollovers, the Baseline period was obtained from the core studies of EP0083 and N01358 directly. A negative value in percent change from Baseline indicates a decrease in PSF from Baseline. Evaluation Period values for seizure frequency were calculated from the seizure diary data collected during the Evaluation Period on/after the first BRV administration.
Time Frame: Baseline of EP0083 or N01358 and up to 84 months of Evaluation Period
Population: The Full Analysis Set (FAS) consisted of all participants who took at least 1 dose of study medication and have at least 1 seizure record on Daily Record Card (DRC) during the Evaluation Period.
Measure: Median (Full Range); unit: percent change
Arm/Group | EP0083 Placebo | EP0083 BRV All | N01379 BRV
Number analyzed (Participants) | 54 | 112 | 7
percent change | 60.6 [-87 to 100] | 43.2 [-497 to 100] | 67.0 [-72 to 100]

3. Secondary Outcome: 50 Percent (%) Responder Rate in Partial Seizure Frequency Per 28 Days From Baseline of EP0083 or N01358 to the Evaluation Period for Rollover Study Participants
Description: The seizure frequency was calculated as number of seizures per 28 days. 50% responders were defined as a participant with a >= 50% reduction in seizure frequency from the baseline period over the post-baseline period. Percentages are based on the number of participants who performed the seizure assessment at each time point. Evaluation Period values for seizure frequency were calculated from the seizure diary data collected during the Evaluation Period on/after the first BRV administration.
Time Frame: Baseline of EP0083 or N01358 and up to 84 months of Evaluation Period
Population: The FAS consisted of all participants who took at least 1 dose of study medication and have at least 1 seizure record on DRC during the Evaluation Period.
Measure: Number; unit: percentage of responders
Arm/Group | EP0083 Placebo | EP0083 BRV All | N01379 BRV
Number analyzed (Participants) | 54 | 112 | 7
percentage of responders | 66.7 | 47.3 | 57.1

4. Secondary Outcome: Percent Change in Partial Seizure Frequency Per 28 Days From Baseline of Directly Enrolled Study Participants to the Evaluation Period
Description: The seizure frequency was calculated as number of seizures per 28 days. For direct enrollers, the Baseline Period was defined as seizure counts collected from 8 weeks prior to the first BRV administration in EP0085. Change in seizure frequency is calculated as the seizure frequency at the evaluation time point minus the seizure frequency at Baseline of directly enrolled participants. A negative value in percent change from Baseline indicates a decrease in PSF from Baseline. Evaluation Period values for seizure frequency were calculated from the seizure diary data collected during the Evaluation Period on/after the first BRV administration.
Time Frame: Baseline (8 weeks prior to BRV administration), up to 39 months of Evaluation Period
Population: as for outcome 3
Measure: Median (Full Range); unit: percent change
Arm/Group | Direct Enrollers BRV
Number analyzed (Participants) | 34
percent change | -32.6 [-3691 to 100]

5. Secondary Outcome: 50 % Responder Rate in Partial Seizure Frequency Per 28 Days Over the Evaluation Period for Directly Enrolled Study Participants
Description: The seizure frequency for directly enrolled participants was calculated as number of seizures per 28 days from 8 weeks prior to BRV administration. 50% responders were defined as a participant with a >= 50% reduction in seizure frequency from the Baseline Period over the post-baseline period. Percentages are based on the number of participants who performed the seizure assessment at each time point. For direct enrollers, the Baseline Period was defined as seizure counts collected from 8 weeks prior to the first BRV administration in EP0085. Evaluation Period values for seizure frequency were calculated from the seizure diary data collected during the Evaluation Period on/after the first BRV administration.
Time Frame: Baseline (8 weeks prior to BRV administration), up to 39 months of Evaluation Period
Population: as for outcome 3
Measure: Number; unit: percentage of responders
Arm/Group | Direct Enrollers BRV
Number analyzed (Participants) | 34
percentage of responders | 26.5

6. Secondary Outcome: Percentage of Participants Continuously Seizure-free for Partial Seizure and All Seizure Types (Partial, Generalized, and Unclassified Epileptic Seizure) for at Least 6 Months During the Evaluation Period for Rollover Study Participants
Description: A study participant was considered seizure free, if no seizure occurred during 6 consecutive months in the Evaluation Period and if met all of the following criteria: - the participant completed the designated period during the Evaluation Period - the participant has at least 90% non-missing diary days during the period of time - the participant did not report any seizures during the period.
Time Frame: During the Evaluation Period (up to 84 months)
Population: The FAS consisted of all participants who took at least 1 dose of study medication and have at least 1 seizure record on DRC during the Evaluation Period. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | EP0083 Placebo | EP0083 BRV All | N01379 BRV
Number analyzed (Participants) | 52 | 101 | 7
percentage of participants | 15.4 | 19.8 | 28.6

7. Secondary Outcome: Percentage of Participants Continuously Seizure-free for Partial Seizure and All Seizure Types (Partial, Generalized, and Unclassified Epileptic Seizure) for at Least 12 Months During the Evaluation Period for Rollover Study Participants
Description: A study participant was considered seizure free, if no seizure occurred during 12 consecutive months in the Evaluation Period and if met all of the following criteria: - the participant completed the designated period during the Evaluation Period - the participant has at least 90% non-missing diary days during the period of time - the participant did not report any seizures during the period.
Time Frame: During the Evaluation Period (up to 84 months)
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | EP0083 Placebo | EP0083 BRV All | N01379 BRV
Number analyzed (Participants) | 48 | 93 | 6
percentage of participants | 8.3 | 14.0 | 33.3

8. Secondary Outcome: Percentage of Participants Continuously Seizure-free for Partial Seizure and All Seizure Types During the Evaluation Period for Rollover Study Participants
Description: A study participant was considered seizure free (partial, all epileptic seizure), if no seizure occurred during the Evaluation Period and if met all of the following criteria: - the participant completed the designated period during the Evaluation Period - the participant has at least 90% non-missing diary days during the period of time - the participant did not report any seizures during the period.
Time Frame: During the Evaluation Period (up to 84 months)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | EP0083 Placebo | EP0083 BRV All | N01379 BRV
Number analyzed (Participants) | 54 | 112 | 7
percentage of participants
  Participants with partial seizure-freedom | 1.9 | 7.1 | 14.3
  Participants with all-type seizure-freedom | 1.9 | 7.1 | 14.3

9. Secondary Outcome: Percentage of Participants Continuously Seizure-free for Partial Seizure and All Seizure Types (Partial, Generalized, and Unclassified Epileptic Seizure) for at Least 6 Months During the Evaluation Period for Directly Enrolled Study Participants
Description: as for outcome 6
Time Frame: During the Evaluation Period (up to 39 months)
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Direct Enrollers BRV
Number analyzed (Participants) | 29
percentage of participants | 24.1

10. Secondary Outcome: Percentage of Participants Continuously Seizure-free for Partial Seizure and All Seizure Types (Partial, Generalized, and Unclassified Epileptic Seizure) for at Least 12 Months During the Evaluation Period for Directly Enrolled Study Participants
Description: as for outcome 7
Time Frame: During the Evaluation Period (up to 39 months)
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Direct Enrollers BRV
Number analyzed (Participants) | 26
percentage of participants | 15.4

11. Secondary Outcome: Percentage of Participants Continuously Seizure-free for Partial Seizure and All Seizure Types During the Evaluation Period for Directly Enrolled Study Participants
Description: as for outcome 8
Time Frame: During the Evaluation Period (up to 39 months)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Direct Enrollers BRV
Number analyzed (Participants) | 34
percentage of participants
  Participants with partial seizure-freedom | 5.9
  Participants with all-type seizure-freedom | 5.9

ADVERSE EVENTS:
Time Frame: From Baseline until end of the safety follow up (up to 88.5 months)
Description: Treatment-emergent AEs (TEAEs) were defined as AEs that had onset on or after the day of first BRV dose in EP0085 study. The Safety Set consisted of all participants who took at least 1 dose of study medication.
Arm/Group | EP0083 Placebo | EP0083 BRV All | N01379 BRV | Direct Enrollers BRV
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/112 | 0/7 | 0/34
Serious Adverse Events (participants affected / at risk) | 6/54 | 23/112 | 5/7 | 6/34
Other Adverse Events (participants affected / at risk) | 41/54 | 87/112 | 6/7 | 27/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EP0083 Placebo (N=54) | EP0083 BRV All (N=112) | N01379 BRV (N=7) | Direct Enrollers BRV (N=34)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericoronitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pilonidal cyst (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scapula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian clear cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parkinsonism (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure cluster (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Mental disorder due to a general medical condition (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Self injurious behaviour (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Brain operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Abortion induced (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cranioplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vagal nerve stimulator implantation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EP0083 Placebo (N=54) | EP0083 BRV All (N=112) | N01379 BRV (N=7) | Direct Enrollers BRV (N=34)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 14 (20) | 0 (0) | 4 (4)
Nausea (Gastrointestinal disorders) | 5 (7) | 11 (13) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 3 (6) | 6 (6) | 0 (0) | 3 (6)
Abdominal pain (Gastrointestinal disorders) | 3 (5) | 6 (8) | 1 (2) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 2 (3) | 6 (9) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 5 (6) | 5 (5) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 4 (11) | 4 (4) | 0 (0) | 3 (5)
Pyrexia (General disorders) | 9 (14) | 21 (43) | 1 (2) | 6 (7)
Corona virus infection (Infections and infestations) | 13 (13) | 32 (34) | 0 (0) | 11 (11)
Nasopharyngitis (Infections and infestations) | 20 (88) | 18 (68) | 3 (6) | 9 (19)
Upper respiratory tract infection (Infections and infestations) | 5 (11) | 23 (36) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 3 (3) | 5 (7) | 0 (0) | 3 (13)
Contusion (Injury, poisoning and procedural complications) | 7 (8) | 11 (19) | 2 (10) | 4 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (9) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 8 (12) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 12 (13) | 17 (21) | 3 (4) | 5 (5)
Headache (Nervous system disorders) | 10 (17) | 21 (30) | 0 (0) | 3 (8)
Somnolence (Nervous system disorders) | 14 (17) | 8 (13) | 2 (2) | 6 (8)
Insomnia (Psychiatric disorders) | 5 (6) | 7 (7) | 1 (1) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (12) | 11 (19) | 1 (1) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 13 (17) | 0 (0) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 4 (10) | 7 (11) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/77/NCT03250377/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-03): https://cdn.clinicaltrials.gov/large-docs/77/NCT03250377/SAP_001.pdf